CLINICAL TRIAL: NCT02543294
Title: REcovery of Left Ventricular Dysfunction in CAncer Patients (RECAP Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0379
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure; Cancer Treatment Induced Left Ventricular Dysfunction
Keywords: Heart Failure; Echocardiogram; ECHO; Electrocardiogram; ECG; Questionnaire; Survey; Telephone Follow-Up; HF; Cancer treatment induced left ventricular dysfunction; CILVD; Left ventricular ejection fraction; LVEF
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography; Electrocardiography; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anthracycline Treatment Group (Experimental): Participants undergo echocardiograms with contrast done at baseline and at months 2, 4, 6, 12, 18, and 30. Electrocardiogram performed at baseline. Symptom questionnaire completed at baseline and at months 1, 2, 4, 6, 12, 18, and 30. Telephone follow-up by study staff at months 3 and 5.
  Interventions: Device: Echocardiograms; Device: Electrocardiogram; Behavioral: Symptom Questionnaire; Behavioral: Telephone Follow-Up
- Herceptin Treatment Group (Experimental): Participants undergo echocardiograms with contrast done at baseline and at months 2, 4, 6, 12, 18, and 30. Electrocardiogram performed at baseline. Symptom questionnaire completed at baseline and at months 1, 2, 4, 6, 12, 18, and 30. Telephone follow-up by study staff at months 3 and 5.
  Interventions: Device: Echocardiograms; Device: Electrocardiogram; Behavioral: Symptom Questionnaire; Behavioral: Telephone Follow-Up
- Combination of Treatments Group (Experimental): Participants undergo echocardiograms with contrast done at baseline and at months 2, 4, 6, 12, 18, and 30. Electrocardiogram performed at baseline. Symptom questionnaire completed at baseline and at months 1, 2, 4, 6, 12, 18, and 30. Telephone follow-up by study staff at months 3 and 5.
  Interventions: Device: Echocardiograms; Device: Electrocardiogram; Behavioral: Symptom Questionnaire; Behavioral: Telephone Follow-Up

INTERVENTIONS:
Device: Echocardiograms — Participants undergo echocardiograms with contrast done at baseline and at months 2, 4, 6, 12, 18, and 30.
  Other Names: ECHO
Device: Electrocardiogram — Electrocardiogram performed at baseline.
  Other Names: ECG
Behavioral: Symptom Questionnaire — Symptom questionnaire completed at baseline and at months 1, 2, 4, 6, 12, 18, and 30.
  Other Names: Survey
Behavioral: Telephone Follow-Up — Telephone follow-up by study staff at months 3 and 5.

SUMMARY:
The goal of this clinical trial is to learn if heart function remains normal after stopping heart failure medication in patients who have received chemotherapy.

DETAILED DESCRIPTION:
If you agree to take part in this study, the following baseline tests and procedures will be performed on Day 1:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, and breathing rate).
* You will complete a questionnaire about any symptoms you may be having. The questionnaire should take about 5-10 minutes to complete.
* You will have an echocardiogram (ECHO) and an electrocardiogram (ECG) to check your heart function.
* You will have blood (about 3 tablespoons) drawn for routine tests. If you can become pregnant, part of this blood draw will be used for a pregnancy test. To take part in this study, you must not be pregnant.
* You will be given instructions on how to gradually wean yourself off of your heart failure medication.
* You will be given a machine that you will use to measure your blood pressure at home.

You will be asked to monitor your blood pressure and heart rate at home daily and keep the results in a diary. You should bring your diary to each study visit.

At Month 1:

* You will have a physical exam, including measurement of your vital signs.
* You will complete the questionnaire about any symptoms you may be having.
* You will have blood (about 2 teaspoons) drawn for routine tests.

At Months 2, 4, 6, 12, 18, and 30:

* You will have a physical exam, including measurement of your vital signs.
* You will complete the questionnaire about any symptoms you may be having.
* You will have an ECHO.
* You will have blood (about 2 teaspoons) drawn for routine tests.

At Months 3 and 5, you will have a telephone follow-up with a member of the research team.

Length of Study Participation:

You may continue taking part in the study for up to 6 continuous months with follow-up visits at Months 12, 18, and 30. You will no longer be able to take part if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study.

Up to 45 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer survivors with no evidence of disease for at least 6 months as determined by the oncologist and no longer receiving cancer treatment.
2. Prior diagnosis of CILVD with recovered LVEF (i.e. improved to > 50%) for at least 6 months with recommended HF medications (ACE-I or ARB and/or B-blocker).
3. Absence of other causes of cardiomyopathy (e.g. ischemia, hypertension, amyloidosis, or hemochromatosis) per chart review of the clinician's documentation
4. Documented normal LVEF for at least 6 months after the initiation of recommended HF therapy.
5. Age 18 - 80 years. HF clinical guidelines is supported by evidenced-based data from clinical trials which includes individuals up to 80 years of age.
6. Residence within the United States.
7. Ability to read and write English, because the MD Anderson Symptom Inventory -Heart Failure (MDASI-HF) instrument (Fadol et al., 2008) has been validated in English only.

Exclusion Criteria:

1. Participants will be excluded if they have a recurrence that requires anti-cancer treatment.
2. Have a documented history of hypertension, coronary artery disease, myocardial infarction, diabetes mellitus, amyloidosis or hemochromatosis.
3. Exhibiting HF symptoms (e.g. shortness of breath, edema).
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09-10 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anecita Fadol, PHD, MSN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified in the Cardiology outpatient clinic at MD Anderson Cancer Center by research team. Team reviewed cardiac medications (angiotensin-converting-enzyme inhibitor (ACE-I), angiotensin II receptor blocker (ARB), and beta blocker), met with eligible patients, explained study, obtained informed consent, and enrolled in the study.
Groups:
- Intervention (Weaning): Down titrated current dose by half each week until medication is off. Weaning order: ACE-I, ARB, and beta blocker.
Period: Overall Study
Arm/Group | Intervention (Weaning)
Started | 20
Completed | 8
Not Completed | 12
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Patients at MD Anderson that met inclusion criteria (specified in Recruitment Details) and not excluded due to: Cancer recurrence; documented history of hypertension, coronary artery disease, myocardial infarction, diabetes mellitus, amyloidosis or hemochromatosis; presence of HF symptoms (e.g. shortness of breath, edema); Pregnancy.
Arm/Group | Intervention (Weaning)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants] — Maintenance of LVEF ≥50% after weaning of heart failure medications.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 19
    >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (12)
Age, Customized [Count of Participants; unit: Participants]
  < 30 | 1
  >/= 30-39 | 6
  >/= 40-49 | 3
  >/= 50-59 | 6
  >/= 60 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Left ventricular ejection fraction (LVEF) ≥50% [Count of Participants; unit: Participants] — LVEF ≥50%, taking heart failure medications classified as Angiotension converting enzyme inhibitors (ACE-Inhibitors), Beta-blockers, and/or angiotension-receptor blockers (ARBs), no diabetes, no hypertension, no arrhythmias, cancer in remission for at least 6 months
  Participants | 20

OUTCOME MEASURES:

1. Primary Outcome: Determine the Percentage of Cancer Survivors That Maintain Left Ventricular Ejection Fraction (LVEF) ≥50% After Discontinuing Cardiac Medications: Beta Blockers, Angiotensin Converting Enzyme Inhibitors (ACE-I), or Angiotensin Receptor Blockers (ARB).
Description: A withdrawal failure is defined as a decrease in the LVEF when cardiac medications are discontinued as determined by echocardiogram to LVEF<50% or a decrease by 10% from baseline measurement. Maintenance of LVEF is defined as LVEF≥50%. LVEF was assessed at Baseline, Months 2, 4, 6, 12, 18, & 30.
Time Frame: A total of 30 months from enrollment date of each participant;
Measure: Count of Participants; unit: Participants
Groups:
- Intervention (Weaning): "Weaning of Cardiac Medications Based on Therapeutic Category (i.e. Beta Blockers, ACE-I, ARB, or any combination of these medications.)"
Arm/Group | Intervention (Weaning)
Number analyzed (Participants) | 20
Participants
  Maintained (LVEF </= 50%) | 8
  Withdrawal Failure (LVEF <50% or decrease of 10%) | 2
  Lost to Follow Up | 3
  Withdrawal by Subject | 7

2. Secondary Outcome: Risk Factors to Predict Early Decline of Myocardial Function During the Weaning of HF (Heart Failure) Medications.
Description: To identify an increased troponin-I that can predict the possibility of HF medication withdrawal failure.
Time Frame: A total of 30 months from enrollment date of each participant
Population: The standard deviation is 0 because every value collected over the course of the entire study was 0.03. Mean would be 0.03 with a standard deviation of 0
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Intervention (Weaning)
Number analyzed (Participants) | 20
ng/mL | 0.03 (0)

ADVERSE EVENTS:
Time Frame: Thirty (30) months from date of enrollment
Groups:
- Intervention (Weaning): Weaning of Cardiac Medications Based on Therapeutic Category (i.e. Beta Blockers, ACE-I, ARB, or any combination of these medications.)
Arm/Group | Intervention (Weaning)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (Weaning) (N=20)
Decrease in Ejection fraction (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT02543294/Prot_SAP_000.pdf